CLINICAL TRIAL: NCT01087931
Title: Local Anesthetic Use at Iliac Crest Bone Graft Site in Spinal Reconstructive Surgery
Brief Title: Pain Relief at Iliac Crest Bone Harvest Sites in Spine Surgery Using Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 100096
Record Dates: First submitted 2010-03-11; First posted 2010-03-16 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Local anesthetic; Iliac crest bone harvest; Patients undergoing spine surgery that require use of iliac crest bone autograft
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): This group will receive bupivacaine (10ml of 0.5%) administered directly into the surgical wound at the iliac crest bone harvest site.
  Interventions: Drug: Bupivacaine
- Saline (Placebo Comparator): This group will receive normal saline (10ml) administered directly into the surgical wound at the iliac crest bone harvest site.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine — Single application of 10ml of bupivacaine 0.5% into the iliac crest bone harvest surgical site.
  Other Names: Marcaine.
  Arms: Bupivacaine
Other: Normal Saline — Normal saline 0.9%, 10ml, single application directly into iliac crest bone harvest surgical site.
  Arms: Saline

SUMMARY:
The use of iliac crest bone graft (ICBG) remains the gold-standard in spinal reconstructive surgery for achieving fusion. Major complications from the harvesting of ICBG are rare, but chronic pain has been reported in 10-39%. Catheters implanted at the time of surgery have been used to provide local anesthetic at the harvest site for 24-48 hours after surgery. This has been shown to decrease chronic pain at 4 years post-operatively. A single application of local anesthetic at surgery has been shown to decrease pain at the harvest site for up to 5 days. No study has demonstrated a benefit to using a single application of local anesthetic at the ICBG site beyond 5 days. In current clinical practice, the use of a local anesthetic at the ICBG site is determined according to surgeon preference. The purpose of this study is to determine if a single application of bupivacaine at the ICBG site, as currently done in some cases, provides any pain relief beyond 5 days such as that demonstrated with longer infusions of local anesthetics.

DETAILED DESCRIPTION:
The use of local anesthetic at the donor site has been investigated to decrease the morbidity of iliac crest bone harvesting. Along with a decrease in early post-operative pain that may be expected a decrease in chronic pain and improved long-term results have also been demonstrated. Local anesthetics may cause such long-term results by dampening the initial chemical response to injury by reducing the release of inflammatory mediators from neutrophils, neutrophil adhesion to the endothelium, and the formation of free oxygen radicals. Most studies have utilized continuous or periodic infusions of anesthetic through a catheter placed at the time of surgery for 24-48 hours postoperatively. The drawbacks to using a catheter include increased infection risk and increased cost if a continuous infusion is used . A single treatment of local anesthetic at the time of surgery is therefore preferable. Only one study has evaluated a single injection of local anesthetic in adult spine patients, demonstrating decreased pain and narcotic usage through 5 post-operative days. No study to date has demonstrated a decrease in intermediate or long-term donor site pain through a single application of anesthetic, as achieved in previous studies utilizing post-operative infusions via a catheter.

Participants in the study will be identified in by the attending surgeons on this study who are clinical faculty within the department of orthopaedics and board certified in spine surgery. Randomization will be done by random selection of a sealed envelope by the attending physician at the time of enrollment. Sealed envelopes will contain a paper that assigns the patient to the treatment (bupivacaine at bone harvest site) or placebo (normal saline at bone harvest site) group. Note that all surgical wounds are routinely irrigated with normal saline prior to skin closure. In the control group, 10ml more of normal saline will be used in the ICBG site. In the treatment group, 10ml of bupivacaine 0.5% will be administered directly into the surgical wound, as done in some cases currently. Therefore, there are no new procedures in this protocol outside of what is already being done in practice. The current practice of using versus not using local anesthetic at the iliac crest bone graft site is at the discretion of the attending surgeon. Please note that the randomization in this study has nothing to do with the surgery that is done, and all patients will be treated according to standard of care regardless of this randomization. There are no other differences between treatments in the two study groups. There are no deviations from normal post-operative care received.

Patients will not be told whether or not they receive bupivacaine at the iliac crest bone graft site at the time of surgery. The patient will be blinded to their treatment group throughout the study. At the patient's request, they will be informed of their treatment group at the end of the study. The attending surgeon will not be blinded to the treatment group. The PI will not be blinded to the treatment group.

Background information about the patient and a pain assessment will be done at the time of enrollment by asking participants to fill out a paper questionnaire. Paper questionnaires to assess the patient's pain level will be given to and collected from patients at discharge from the hospital, the first follow up appointment (approximately 2-4 weeks postoperatively), and at the next follow up appointment (approximately 3 months postoperatively). In addition, patients will be given a paper narcotics log to enter their daily oral narcotic usage between the time of discharge and their first follow up appointment.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older undergoing posterior cervical, thoracic, or lumbar surgery
* willingness to participate in the study.

Exclusion Criteria:

* individuals who underwent surgical intervention in the past 6 months
* previous iliac crest bone harvesting
* history of tumor and spondyloarthropathies (rheumatoid arthritis, seronegative arthritis)
* history of adverse reaction to local anesthetic
* history of severe pelvic and hip conditions that can interfere with the outcome assessment of the study
* opioid addiction
* pregnancy
* acute mental illness
* uncontrolled major depression and any other psychiatric disorders
* prisoners
* non-english speaking patients
* inability to understand the informed consent and demands of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R O'Neill, MD, MS, Principal Investigator — Vanderbilt University Medical Center, Department or Orthopaedics; Richard A Davis, MD, Study Chair — Vanderbilt University Medical Center, Department or Orthopaedics; Clint Devin, MD, Study Chair — Vanderbilt University Medical Center, Department or Orthopaedics
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] O'Neill KR, Lockney DT, Bible JE, Crosby CG, Devin CJ. Bupivacaine for pain reduction after iliac crest bone graft harvest. Orthopedics. 2014 May;37(5):e428-34. doi: 10.3928/01477447-20140430-52. PMID 24810818

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine | Saline
Started | 20 | 20
1st Follow up | 20 | 19
Final Follow up | 19 | 17
Completed (all participants completed either the 1st follow-up evaluation or the final evaluation) | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Saline | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 62 (8) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Pain, Cumulative Visual Analog Score, 1st Follow Up
Description: Cumulative Visual Analog Score pain score scores were calculated using the sum of scores (at rest and with movement, pain on average at rest and with movement, and maximum pain at rest and with movement) Range = 0-60 for cumulative visual analog pain score with 0=no pain and 60=worst pain ever.
Time Frame: about 4 to 5 weeks after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine | Saline
Number analyzed (Participants) | 20 | 19
units on a scale | 10.5 (11) | 21.7 (17)

2. Primary Outcome: Pain, Cumulative Visual Analog Score, Final Follow up
Description: as for outcome 1
Time Frame: about 18 to 20 weeks after surgery
Population: Original study data has been lost. Estimated values obtained from a figure describing the results in the study results publication are reported in the data table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine | Saline
Number analyzed (Participants) | 20 | 19
units on a scale | 15.33 (5.55) | 29.33 (7.11)

3. Secondary Outcome: Narcotic Use, 1st Follow up
Description: Number of participants using narcotics for pain
Time Frame: about 4 to 5 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Saline
Number analyzed (Participants) | 20 | 19
Participants | 9 | 13

4. Secondary Outcome: Narcotic Use, Final Follow up
Description: Number of participants using narcotics for pain
Time Frame: about 18 to 20 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Saline
Number analyzed (Participants) | 19 | 17
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Original study data is lost. Adverse event data was pulled from publication based on study.
Arm/Group | Bupivacaine | Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine (N=20) | Saline (N=20)
Superficial Infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Original Study data cannot be found. Data for this record was pulled from the publication, Bupivacaine for pain reduction after iliac crest bone graft harvest, PMID: 24810818.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes